CLINICAL TRIAL: NCT04484935
Title: A Phase 2, Open-label, Uncontrolled, Single-dose Study to Evaluate the Safety and Tolerability, Pharmacokinetics, and Occurrence of Antidrug Antibody for Nirsevimab in Immunocompromised Children ≤ 24 Months of Age
Brief Title: Evaluate the Safety and Tolerability, for Nirsevimab in Immunocompromised Children
Acronym: MUSIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: D5290C00008; 2021-003221-30 (EudraCT Number)
Record Dates: First submitted 2020-06-30; First posted 2020-07-24 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: RSV Infection
Keywords: LRTI by RSV infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — nirsevimab

STUDY DESIGN:
Masking Description: Open: no masking is used. All involved know the identity of the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nirsevimab (Experimental): 1st RSV season: 50mg nirsevimab
  1. st RSV season: 100mg nirsevimab
  2. nd RSV season: 200mg nirsevimab
  Interventions: Drug: Nirsevimab

INTERVENTIONS:
Drug: Nirsevimab — Single fixed IM dose of nirsevimab 50 mg if body weight < 5 kg or 100 mg if body weight ≥ 5 kg, and subjects entering their second RSV season will receive a single fixed IM dose of nirsevimab 200 mg
  Other Names: Nirsevimab (MEDI8897)

SUMMARY:
Study D5290C00008 is a Phase 2, open-label, uncontrolled, single-dose study to evaluate the safety and tolerability, pharmacokinetic(s) (PK), occurrence of antidrug antibody (ADA), and efficacy of nirsevimab in immunocompromised children who are ≤ 24 months of age at the time of dose administration. Approximately 100 subjects will be enrolled. Subjects will be followed for approximately 1 year after dose administration.

DETAILED DESCRIPTION:
Respiratory syncytial virus (RSV) is the most common cause of lower respiratory tract infection (LRTI) among infants and young children, resulting in annual epidemics in Japan. Children with congenital or acquired immunodeficiencies, transplant recipients, and those receiving immunosuppressive therapy are at increased risk for severe RSV-associated LRTI with prolonged viral shedding and higher viral loads, resulting in prolonged hospitalizations, admissions to the intensive care unit (ICU), and the need for mechanical ventilation. Palivizumab (Synagis®) is the only approved agent for RSV prophylaxis, and its half-life (t1/2) is approximately 1 month, infants and young children need to receive monthly intramuscular doses of palivizumab throughout the RSV season to maintain protection. This constitutes a significant burden on healthcare providers as well as the infants/children and their families.

Nirsevimab may provide a cost-effective opportunity to protect all infants from RSV disease based on an improvement in potency and the extended t1/2 that is expected to support once-per-RSV-season dosing.

ELIGIBILITY:
Inclusion Criteria:

* Neonate, infant, or young child ≤ 24 months of age at the time of dose administration who, per investigator judgement, are:

  1. In their first year of life AND entering their first RSV season at the time of dose administration OR
  2. In their second year of life AND entering their second RSV season at the time of dose administration
* The subject must meet at least 1 of the following conditions at the time of informed consent.

  1. Diagnosed with combined immunodeficiency (severe combined immunodeficiency, X-linked hyper-immunoglobulin M [IgM] syndrome, etc); antibody deficiency (X linked agammaglobulinemia, common variable immunodeficiency, non-X-linked hyper-IgM syndromes, etc); or other immunodeficiency (Wiskott-Aldrich syndrome, DiGeorge syndrome, etc), or
  2. Diagnosed with human immunodeficiency virus infection, or
  3. History of organ or bone marrow transplantation, or
  4. Subject is receiving immunosuppressive chemotherapy, or
  5. Subject is receiving systemic high-dose corticosteroid therapy (prednisone equivalents ≥ 0.5 mg/kg every other day, other than inhaler or topical use), or
  6. Subject is receiving other immunosuppressive therapy (eg, azathioprine, methotrexate, mizoribine, mycophenolate mofetil, cyclophosphamide, cyclosporine, tacrolimus, cytokine inhibitors, etc)
* Written informed consent and any locally required authorization obtained from the subject's parent(s)/legal representative(s) prior to performing any protocol-related procedures, including screening evaluations.
* Subject's parent(s)/legal representative(s) able to understand and comply with the requirements of the protocol including follow-up visits as judged by the investigator.
* Subject is available to complete the follow-up period, which will be approximately 1 year after receipt of nirsevimab

Exclusion Criteria:

* Subject who meets any of the palivizumab indications approved in Japan other than immunocompromised condition.

  1. Subject born at ≤ 28 weeks gestation and is ≤ 12 months of age
  2. Subject born at 29 to 35 weeks gestation and is ≤ 6 months of age
  3. Age ≤ 24 months with a history of bronchopulmonary dysplasia requiring medical management within the past 6 months
  4. Age ≤ 24 months with current hemodynamically significant congenital heart disease (CHD)
  5. Age ≤ 24 months with Down syndrome
* Requirement for oxygen supplementation, mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure, or other mechanical respiratory or cardiac support at screening
* A current, active infection, including RSV infection, at the time of screening or at the time of investigational product administration.
* Any fever (≥ 100.4°F [≥ 38.0°C], regardless of route) or acute illness within 7 days prior to investigational product administration.
* Any serious concurrent medical condition (renal failure, hepatic dysfunction, suspected active or chronic hepatitis infection, seizure disorder, unstable neurologic disorder, etc), except those resulting in an immune deficiency condition.
* Clinically significant congenital anomaly of the respiratory tract.
* Receipt of palivizumab.
* Any known allergy or history of allergic reaction to any component of nirsevimab.
* Any known allergy or history of allergic reaction to immunoglobulin products, blood products, or other foreign proteins.
* Concurrent enrollment in another interventional study, or prior receipt of any investigational agent.
* Anticipated survival of less than 1 year at the time of informed consent.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of study results.
* Children of employees of the sponsor, clinical study site, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Tampa, Florida
  - Research Site, Syracuse, New York
  - Research Site, North Charleston, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Tacoma, Washington
- Belgium (2):
  - Research Site, Brussels
  - Research Site, Liège
- Japan (9):
  - Research Site, Bunkyō City
  - Research Site, Fuchu-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Nagasaki
  - Research Site, Setagaya-ku
  - Research Site, Tsukuba
  - Research Site, Yokohama
- Research Site, Bydgoszcz, Poland
- South Africa (2):
  - Research Site, Parktown
  - Research Site, Soweto
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
- Ukraine (2):
  - Research Site, Dnipro
  - Research Site, Kharkiv
- Research Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AstraZeneca (AZ) disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AstraZeneca (AZ) are accepting requests for Individual Participant Data (IPD), but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the European Federation of Pharmaceutical Industries and Associations (EFPIA) Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSRsynopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00008&attachmentIdentifier=e1f614d0-cc7a-48b9-bd02-b07ef3f57993&fileName=D5290C00008_(MUSIC)_CSR_synopsis_Redacted_PDFA.pdf&versionIdentifier=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00008&attachmentIdentifier=f452db79-fd73-45bd-9478-ced954a3eb54&fileName=D5290C00008_(MUSIC)_CSP_V3_Redacted_PDFA.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00008&attachmentIdentifier=1090bbf3-81c1-4d00-817c-6702bdc5ae4d&fileName=D5290C00008_(MUSIC)_SAP_ed-3_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2, open-label, uncontrolled, single-dose study was conducted at 28 investigational sites in 8 countries (Belgium, Japan, Poland, South Africa, Spain, Ukraine, United Kingdom and United States) in immunocompromised children who were <=24 months of age at the time of enrollment between 19 Aug 2020 and 17 Feb 2023.
Pre-assignment Details: This study consisted of a screening period (Visit 1, Day -30 to Day -1); a dosing visit (Visit 2, Day 1) where participants received treatment with nirsevimab and a follow-up period up to Day 361 (Visit 3 to 7). A total of 100 children were enrolled in this study.
Groups:
- Nirsevimab 50 mg/100 mg: Participants in their first year of life with a body weight <5 kilograms (kg) received a single fixed intramuscular (IM) dose of 50 milligram (mg) nirsevimab and those with body weight >=5 kg received a single fixed IM dose of 100 mg nirsevimab.
- Nirsevimab 200 mg: Participants in their second year of life received a single fixed IM dose of 200 mg (2 × 100 mg) of nirsevimab.
Period: Overall Study
Arm/Group | Nirsevimab 50 mg/100 mg | Nirsevimab 200 mg
Started | 48 | 52
Completed | 45 | 49
Not Completed | 3 | 3
Not completed — Other | 0 | 1
Not completed — Withdrawal by parent/guardian | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Population: The As-treated population consisted of all participants who were enrolled and received any dose of nirsevimab.
Groups:
- Nirsevimab 50 mg/100 mg: Participants in their first year of life with a body weight <5 kg received a single fixed IM dose of 50 mg nirsevimab and those with body weight >=5 kg received a single fixed IM dose of 100 mg nirsevimab.
- Total: Total of all reporting groups
Arm/Group | Nirsevimab 50 mg/100 mg | Nirsevimab 200 mg | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.64 (3.270) | 17.90 (3.748) | 12.97 (6.232)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 30 | 35 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 44 | 49 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 16 | 12 | 28
  American Indian or Alaskan Native | 1 | 0 | 1
  Black or African American | 9 | 11 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 20 | 25 | 45
  Other | 2 | 2 | 4
  Multiple categories checked | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious AEs (TESAEs), AEs of Special Interest (AESIs), and New Onset Chronic Disease (NOCDs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the treatment. TEAEs were AEs whose onset occurred after receiving nirsevimab and within 360 days post dose. A TESAE was any AE that resulted in death, was life-threatening, required inpatient hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality, or was medically significant. AESIs were defined as AEs of immediate (type I) hypersensitivity (including anaphylaxis), thrombocytopenia, and immune complex disease following the administration of nirsevimab based on investigator assessment and Medical Dictionary for Regulatory Activities (MedDRA) preferred term (PT) codes. An NOCD was a newly diagnosed medical condition of a chronic, ongoing nature post administration of treatment.
Time Frame: TEAEs were collected from the first dose administration (Day 1) up to 360 days post dose
Population: The As-treated population consisted of all participants who were enrolled and received any dose of nirsevimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab 50 mg/100 mg | Nirsevimab 200 mg
Number analyzed (Participants) | 48 | 52
Participants
  Any TEAE | 36 | 45
  TESAE | 12 | 20
  AESI based on investigator assessment | 3 | 2
  AESI based on selected MedDRA PT codes | 16 | 13
  NOCD | 0 | 0

2. Secondary Outcome: Serum Concentrations of Nirsevimab
Description: Serum concentrations of nirsevimab at selected time points were evaluated to confirm that adequate exposures for protection from respiratory syncytial virus (RSV) lower respiratory tract infection (LRTI) are maintained for at least 5 months after dosing.
Time Frame: Baseline (Day 1) and on Days 8 (for Japanese participants), 31, 151 and 361
Population: The As-treated population consisted of all participants who were enrolled and received any dose of nirsevimab. Only those participants with data available are included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Nirsevimab 50 mg/100 mg | Nirsevimab 200 mg
Number analyzed (Participants) | 48 | 52
mcg/mL
  Baseline (Day 1) | NA (NA) — Data was below the lower limit of quantification [0.5 microgram (mcg)/mL] | NA (NA) — Data was below the lower limit of quantification (0.5 mcg/mL)
  Day 8: number analyzed (Participants) | 15 | 11
  Day 8 | 139.24 (22.26) | 206.79 (16.58)
  Day 31: number analyzed (Participants) | 47 | 50
  Day 31 | 66.00 (141.06) | 109.77 (91.74)
  Day 151: number analyzed (Participants) | 39 | 44
  Day 151 | 19.80 (101.19) | 24.14 (121.54)
  Day 361: number analyzed (Participants) | 29 | 38
  Day 361 | 1.86 (119.96) | 1.93 (158.95)

3. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Nirsevimab
Description: Blood samples were analyzed for the presence of ADAs for nirsevimab using validated assays.
Time Frame: Baseline (Day 1) and on Days 31, 151 and 361
Population: The As-treated population consisted of all participants who were enrolled and received any dose of nirsevimab. Only those participants with data available were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab 50 mg/100 mg | Nirsevimab 200 mg
Number analyzed (Participants) | 48 | 52
Participants
  Day 1 | 0 | 0
  Day 31 | 0 | 1
  Day 151 | 1 | 0
  Day 361 | 2 | 7

4. Secondary Outcome: Number of Participants With Medically Attended (MA) RSV LRTI (Inpatient and Outpatient) and Hospitalizations
Description: Number of participants with LRTI and hospitalizations due to reverse transcriptase-polymerase chain reaction (RT-PCR)-confirmed RSV was assessed. MA RSV LRTI consisted of participants with protocol-defined LRTI, positive central RT-PCR RSV test result, Investigator assessed LRTI at an inpatient or outpatient setting. MA RSV LRTI with hospitalization consisted of participants with protocol-defined LRTI, positive central RT-PCR RSV test result, Investigator assessed LRTI at an inpatient setting.
Time Frame: Through 150 days post dose
Population: The As-treated population consisted of all participants who were enrolled and received any dose of nirsevimab.
Measure: Count of Participants; unit: Participants
Arm/Group | Nirsevimab 50 mg/100 mg | Nirsevimab 200 mg
Number analyzed (Participants) | 48 | 52
Participants
  MA RSV LRTI | 0 | 0
  MA RSV LRTI with hospitalization | 0 | 0

ADVERSE EVENTS:
Time Frame: The TEAEs were collected from the first dose administration (Day 1) up to 360 days post dose
Description: The As-treated population consisted of all participants who were enrolled and received any dose of nirsevimab.
Arm/Group | Nirsevimab 50 mg/100 mg | Nirsevimab 200 mg
All-Cause Mortality (participants affected / at risk) | 2/48 | 1/52
Serious Adverse Events (participants affected / at risk) | 12/48 | 20/52
Other Adverse Events (participants affected / at risk) | 35/48 | 41/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirsevimab 50 mg/100 mg (N=48) | Nirsevimab 200 mg (N=52)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Serratia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrostomy failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sickle cell disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Feeding intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 2 (3)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 3 (3)
Candida sepsis (Infections and infestations) | 2 (2) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (2) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Giardiasis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nirsevimab 50 mg/100 mg (N=48) | Nirsevimab 200 mg (N=52)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (13) | 6 (9)
Otitis media (Infections and infestations) | 5 (7) | 6 (7)
Otitis media acute (Infections and infestations) | 2 (9) | 4 (5)
Rhinitis (Infections and infestations) | 2 (2) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 18 (49) | 18 (33)
Viral upper respiratory tract infection (Infections and infestations) | 4 (7) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 7 (9)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5 (6) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Eczema infantile (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (4) | 2 (4)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 10 (15)
Vomiting (Gastrointestinal disorders) | 8 (13) | 13 (16)
Pyrexia (General disorders) | 13 (25) | 13 (27)
COVID-19 (Infections and infestations) | 4 (4) | 12 (12)
Conjunctivitis (Infections and infestations) | 4 (5) | 2 (3)
Ear infection (Infections and infestations) | 0 (0) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (2) | 6 (7)
Gastroenteritis viral (Infections and infestations) | 3 (5) | 4 (4)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 4 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT04484935/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT04484935/SAP_001.pdf